CLINICAL TRIAL: NCT06597812
Title: The Effect of Two Different Modes of Anaesthesia Mainantance on Postoperative Delirium in Elderly Patient with Low Preoperative Mini-cog Score
Brief Title: The Effect of Two Different Modes of Anaesthesia Mainantance on Postoperative Delirium
Status: Completed | Type: Observational
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Harun Tolga Duran, head of Anaesthesiology and reanimation department, Amasya University
Other Study IDs: 2023/11
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cognitive Dysfunction, Cognitive Disorder; Delirium - Postoperative
Keywords: delirium; Mini-Cog; anaesthesia
MeSH Terms: conditions — Cognitive Dysfunction; Emergence Delirium; Delirium | interventions — Sevoflurane

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- group s: Patients receiving sevoflurane
  Interventions: Procedure: Sevoflurane
- Group p: Patients receiving propofol-based total intravenous anesthesia
  Interventions: Procedure: Sevoflurane

INTERVENTIONS:
Procedure: Sevoflurane — Depending on the anesthesia maintenance protocol, total intravenous anesthesia (TIVA) or sevoflurane anesthesia, patients were divided into group T (TIVA) and group S (sevoflurane).

SUMMARY:
In this study, the cognitive status of the patients in the preoperative period was taken into consideration and the development of delirium after the surgery was investigated. There is no harm to the patient.

DETAILED DESCRIPTION:
The patients were preoperatively assessed for American Society of Anesthesiologists (ASA) risk by an anesthetist and age, sex and comorbidities were recorded. The Mini-cog test was applied as a cognitive screening test by the anesthesiologist in the preoperative period and the test score was recorded. Three-word memory test, clock drawing, and visual function test was performed to evaluate the patient's cognitive functions. In this test, patients were asked to memorize three words such as umbrella, sunshine, and chair at the beginning of the test.

ELIGIBILITY:
Inclusion Criteria:

* There was a correlation between the incidence of delirium after the age of 60(10).

Exclusion Criteria:

* Patients' age< 60 years,
* Patients undergoing emergency cholecystectomy or did not have preoperative Mini-Cog assessment,
* With a history of cerebrovaskuler insult that was thought to have an effect on postoperative delirium ,
* Patients with difficulty in cooperation ,
* Patients with hemodynamic instability(arterial blood pressure above 160/90 mmHg and below 90/60 mmHg and patients with pulse rate below 50/min and above 100/min) ,
* Patients with previously diagnosed dementia, and those who had surgical procedures lasting more than 2 hours were excluded from the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over 60 years of age who are scheduled for laparoscopic cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Group P-S | postoperative 0 1st 2nd hours
  Incidence of postoperative delirium in patients receiving sevoflurane or propofol-based total intravenous anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya University Hospital, Amasya, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I approve the usability in multicenter studies in the study plan population

REFERENCES:
- [Background] Fiamanya S, Ma S, Yates DRA. The association between preoperative Mini-Cog(c) score and postoperative delirium (POD): a retrospective cohort study. Perioper Med (Lond). 2022 Apr 21;11(1):16. doi: 10.1186/s13741-022-00249-0. PMID 35443735
- [Background] Jing GW, Xie Q, Tong J, Liu LZ, Jiang X, Si L. Early Intervention of Perioperative Delirium in Older Patients (>60 years) with Hip Fracture: A Randomized Controlled Study. Orthop Surg. 2022 May;14(5):885-891. doi: 10.1111/os.13244. Epub 2022 Apr 19. PMID 35441485
- [Background] Racine AM, Fong TG, Gou Y, Travison TG, Tommet D, Erickson K, Jones RN, Dickerson BC, Metzger E, Marcantonio ER, Schmitt EM, Inouye SK. Clinical outcomes in older surgical patients with mild cognitive impairment. Alzheimers Dement. 2018 May;14(5):590-600. doi: 10.1016/j.jalz.2017.10.010. Epub 2017 Nov 27. PMID 29190460
- [Derived] Duran HT, Kizilkaya M, Aydinli A, Osmantevfik S, Tastan S, Kilinc OO, Pirhan Y. The effect of two different modes of anaesthesia maintenance on postoperative delirium in elderly patient with low preoperative mini-cog score. BMC Anesthesiol. 2024 Oct 1;24(1):350. doi: 10.1186/s12871-024-02735-y. PMID 39354373
- See also: Related Info — https://mini-cog.com